CLINICAL TRIAL: NCT01652755
Title: Use of Cystatin C in Predicting AKI in Patients Undergone Cardiopulmonary Bypass Surgery
Brief Title: Plasma Cystatin C and Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Hongying Ni, Department vice director, Jinhua Central Hospital
Other Study IDs: N-H-Y
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Acute Kidney Injury
Keywords: cystatin C,acute kidney injury,
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI group: patients with AKI after cardiopulmonary bypass surgery
- non-AKI group: patients without AKI during study period

SUMMARY:
To evaluate the utility of plasma cystatin C(pCysC) as a predictive and diagnostic marker of acute kidney injury(AKI) in patients undergone cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
This is a prospective AKI observational study in patients undergone cardiopulmonary bypass surgery. pCysC and plasma creatine will be measured at entry to ICU.AKI was defined as 50% increase in plasma creatine above baseline.The predictive and diagnostic performance of pCysC will be assessed from area under receiver operator characteristic curve(AUC) and odds ratio(OR).

ELIGIBILITY:
Inclusion Criteria:

* patients with CPB and admitted to ICU

Exclusion Criteria:

* patients with the age >80 or <18 years
* with preexisting renal dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergone cardiopulmonary bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Ni, MM, Study Chair — Jinhua Municipal Central Hospital
Locations (1):
- Jinhua central hospital, Jinhua, Zhejiang, China